CLINICAL TRIAL: NCT04119765
Title: Plasma Oxalate in Patient With Short Bowel
Acronym: OXAGO
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL18_0408
Record Dates: First submitted 2019-10-07; First posted 2019-10-08 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Short Bowel Syndrome; Hyperoxaluria; Hyperoxalemia
MeSH Terms: conditions — Short Bowel Syndrome; Hyperoxaluria | interventions — Blood Specimen Collection; Weights and Measures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Blood sampling — blood sampling will be used to perform oxalemia and FGF23 quantitative analysis
Biological: Urine sampling — urine sampling will be used to measure glycolate urinary rate (glycolaturia) and to perform urinary inflammation markers quantitative analysis
Procedure: Pulse Wave Velocity (PWV) measurement — PWV will be measured thank to the Complior® device
Procedure: central pressure measurement — central pressure will be measured thank to the Complior® device

SUMMARY:
Hyperoxaluria due to fat malabsorption is seen in patients suffering from short bowel and can lead to stones and nephrocalcinosis. Not all patients are prone to these renal complications. only urinary oxaluria is measured in practice. Plasma oxalate shouldn't increase theoretically in these patients. However recent report showed an increase of plasma oxalate in patient with enteric hyperoxaluria. The aim of this study is to assess the plasma oxalate distribution in this specific population to have a new tool to predict renal complication of these patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Type II short bowel for more than 6 months
* Affiliated to a social health care

Exclusion Criteria:

* Primary hyperoxaluria
* Other type of short bowel than type II
* Minor patient or major patient protected by the law

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: type II short bowel patient
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2020-02-27 (Actual); Primary Completion 2022-05-04 (Actual); Study Completion 2022-05-04 (Actual)

PRIMARY OUTCOMES:
Plasma oxalate rate (oxalemia) | at inclusion
  this sample measures the plasma oxalate rate

CONTACTS AND LOCATIONS:
Overall Officials: Sandrine Lemoine, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Nephrology Department, Edouard Herriot Hospital, Lyon, France